CLINICAL TRIAL: NCT05263882
Title: A Phase Ⅱ Single-arm, Open-labelled, Multi-center, Clinical Trial of Gemcitabine Combined With Eribulin for the Treatment of Second-line and Above in Patients With Recurrent HER2 Negative Breast Cancer
Brief Title: Gemcitabine Combined With Eribulin Regimen in the Treatment of Second-line Above Recurrent HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Peijian Peng, professor, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.XBZL.002
Record Dates: First submitted 2022-02-16; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: HER2-negative Breast Cancer
MeSH Terms: interventions — eribulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): * Eribulin mesylate injection, specification: 2ml: 1mg/piece. Usage and dosage: 1.4mg/m2, intravenous bolus injection within 2-5 minutes, 21 days as a cycle, once on the 1st and 8th day of each cycle.
  * Gemcitabine hydrochloride for injection, specification: 200mg: 1g/piece. Usage and dosage: administer gemcitabine (1000 mg/m2) intravenously over 30 minutes on the 1st and 8th day of every 21 days treatment cycle.
  * The above combination regimen takes 21 days as a treatment cycle, and the efficacy is evaluated every 2 treatment cycles. The drug is continued until the disease progresses or intolerable adverse reactions occur.
  Interventions: Drug: Gemcitabine combined with eribulin

INTERVENTIONS:
Drug: Gemcitabine combined with eribulin — * Eribulin mesylate injection, specification: 2ml: 1mg/piece. Usage and dosage: 1.4mg/m2, intravenous bolus injection within 2-5 minutes, 21 days as a cycle, once on the 1st and 8th day of each cycle.
  * Gemcitabine hydrochloride for injection, specification: 200mg: 1g/piece. Usage and dosage: administer gemcitabine (1000 mg/m2) intravenously over 30 minutes on the 1st and 8th day of every 21 days treatment cycle.
  * The above combination regimen takes 21 days as a treatment cycle, and the efficacy is evaluated every 2 treatment cycles. The drug is continued until the disease progresses or intolerable adverse reactions occur.

SUMMARY:
This study intends to conduct a single-arm, open-label Phase II multicenter clinical study of gemcitabine combined with eribulin regimen in the treatment of second-line above recurrent HER2-negative breast cancer. Patients with recurrent HER2-negative breast cancer were recruited, and the efficacy and clinical significance of gemcitabine combined with eribulin regimen in the treatment of recurrent HER2-negative breast cancer second-line above was studied.

ELIGIBILITY:
Inclusion criteria

1. Histologically diagnosed histological examination confirmed breast cancer patients with locally advanced or metastatic HER2-negative (expression lack of human epidermal growth factor 2 (HER2) confirmed by central laboratory examination) and unsuitable for surgical treatment;
2. Received first-line or above systemic therapy in the past, with disease progression after the last treatment, and have used anthracyclines and/or taxanes, and currently there is no standard treatment regimen;
3. Must have at least one evaluable lesion according to RRECIST version 1.1 criteria (the longest diameter on spiral CT is at least 10mm, and the longest diameter on ordinary CT is at least 20mm);
4. Female, 18 years old ≤ aged ≤75 years old;
5. ECOG PS 0~2 points;
6. Expected survival period ≥ 3 months;
7. Sufficient blood function: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥ 80×109/L and hemoglobin ≥ 8g/dL;
8. Sufficient liver function: total bilirubin ≤ 1.5 times the upper limit of normal (ULN); AST and ALT ≤ 2.5 times the upper limit of normal (ULN); alkaline phosphatase ≤ 5 times the upper limit of normal (ULN);
9. Sufficient renal function: serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min;
10. The electrocardiogram is basically normal;
11. Women with an intact uterus must have a negative pregnancy test result within 28 days prior to enrollment in the study (unless it has been 24 months of amenorrhea). If the pregnancy test is more than 7 days from the first dose, a urine pregnancy test is required for verification (within 7 days before the first dose);
12. Have not received radiotherapy, chemotherapy, targeted therapy and other treatments within 4 weeks before enrollment;
13. Signed the informed consent.

Exclusion criteria (Subjects can not enter the study if they meet any of the following conditions)

1. Pregnant, lactating women, or female patients who are fertile but not taking contraceptive measures;
2. Existing severe acute infection that has not been controlled; or purulent and chronic infection with persistent wound healing;
3. Patients with original serious heart disease, including: congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina pectoris, myocardial infarction, severe heart valve disease and resistant hypertension;
4. Those with bleeding tendency;
5. Individual with mental disorders/individual who cannot obtain informed consent;
6. Patients who use drugs and alcohol for a long time, which affects the evaluation of the test results;
7. Other conditions in which the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Recent objective efficacy evaluation | 2 years
  In this clinical study, the efficacy evaluation method of RECIST version 1.1 was adopted, and the objective efficacy changes were evaluated according to the changes in the sum of the longest diameters of each target lesion.

SECONDARY OUTCOMES:
Disease progression-free survival | 2 years
  progression-free survival is defined as the time from the date of randomization to any objectively documented tumor progression or patient death. In the event of a patient lost to follow-up, unexplained death or other anti-tumor therapy, the Disease progression-free survival was calculated up to this point.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 Years
  From the time the patient signed the informed consent form and was enrolled in the trial, any adverse medical event that occurred within 1 month after the end of treatment, regardless of whether it was causally related to the trial drug, was judged as an adverse event (AE). AEs were recorded truthfully during the trial, including the occurrence time, severity, duration, measures taken and outcomes of AEs. The investigator should follow up all AEs until symptoms disappear or the condition stabilizes. For SAEs, they should be followed until properly resolved even after the study ends.

IPD SHARING:
Plan to Share IPD: No